CLINICAL TRIAL: NCT06213857
Title: Clinical Study Evaluating the Possible Beneficial Effect of Silymarin in Patients With Ulcerative Colitis
Brief Title: Beneficial Effect of Silymarin in Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmad Almoutaz Ahmad Eltayeb, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Silymarin in UC
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Silymarin; milk-thistle extract; Mesalamine; Azathioprine

STUDY DESIGN:
Intervention Model Description: This is a randomized parallel study that will be conducted on 44 adult patients with Ulcerative Colitis. Patients will be enrolled after obtaining an informed consent from them or their guardians.
  Patients will be recruited from Rajhy Hospital Outpatient Clinics and Health Insurance Outpatient Clinics at Mabarra Hospital in Assiut, Egypt. The patients will be randomized based on hospital admission days into two groups:
  * Group Ⅰ (Control group): 22 patients will receive Mesalamine (2g/day) + Azathioprine (50mg/day) for 3 months.
  * Group Ⅱ (Silymarin group): 22 patients will receive Mesalamine (2g/day) + Azathioprine (50 mg/day) + Silymarin (140 mg/day) for 3 months.
  The primary outcome will be clinical improvement defined as a 2 point or more decrease in the Mayo score from baseline. The secondary outcomes will be the change in the level of fecal calprotectin, superoxide dismutase and TNF-α.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Control group) (Active Comparator): Mesalamine (2g/day) + Azathioprine (50mg/day) for 3 months
  Interventions: Drug: Mesalamine; Drug: Azathioprine
- B (Silymarin group) (Experimental): Mesalamine (2g/day) + Azathioprine (50mg/day) + Silymarin (140mg/day) for 3 months
  Interventions: Dietary Supplement: Silymarin; Drug: Mesalamine; Drug: Azathioprine

INTERVENTIONS:
Dietary Supplement: Silymarin — Silymarin (milk thistle), an extract obtained from Silybum marianum seeds containing a complex of flavonolignans with a potent intracellular antioxidant property. The first usage of Milk thistle was for its hepatoprotective and antioxidant activities, but in the recent years it has been used to control of immune based murine colitis by healing of bowel histology and reduction of bowel inflammatory cytokines especially TNF-α, interleukin-1β (IL-1β), and nuclear factor κB (NF-κB). Silymarin has anti-viral, immunomodulation, anti-inflammatory effects as well as antioxidant properties by scavenging free radicals and increasing the glutathione concentrations, protective and wound healing effects. It increases the gene expression of antioxidant enzymes and the number of the most important protection mechanisms against free-radicals damage containing superoxide dismutase (SOD), glutathione peroxidase (GPX), and catalase.
  Other Names: Milk Thistle
  Arms: B (Silymarin group)
Drug: Mesalamine — A 5-aminosalicylic acid compound used in the treatment of mild to moderate ulcerative colitis, with high rates of efficacy in induction and maintenance of remission.
  Other Names: Mesalazine
Drug: Azathioprine — An immunosuppressive medication that is used for the treatment of inflammatory bowel disease (Crohn's disease and ulcerative colitis). It works by decreasing the activity of the body's immune system so it will not attack itself.
  Other Names: Immuran

SUMMARY:
The goal of this clinical trial is to evaluate the possible beneficial effect of silymarin in Ulcerative Colitis adult patients receiving mesalamine. This is trial that will be conducted on 44 adult patients with Ulcerative Colitis. Patients will be enrolled after obtaining an informed consent from them or their guardians.

Patients will be recruited from Rajhy Hospital Outpatient Clinics and Health Insurance Outpatient Clinics at Mabarra Hospital in Assiut, Egypt. The patients will be randomized based on hospital admission days into two groups:

* Group Ⅰ (Control group): 22 patients will receive Mesalamine (2g/day) + Azathioprine (50mg/day) for 3 months.
* Group Ⅱ (Silymarin group): 22 patients will receive Mesalamine (2g/day) + Azathioprine (50mg/day) + Silymarin (140 mg/day) for 3 months.

The primary outcome will be clinical improvement defined as a 2 point or more decrease in the Mayo score from baseline. The secondary outcomes will be the change in the level of fecal calprotectin, superoxide dismutase and TNF-α.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD), is a debilitating progressive chronic inflammatory disorder of the small intestine and colon characterized by alternative phases of clinical relapse and remission. IBD includes two types, Crohn's Disease (CD) and Ulcerative Colitis (UC), CD can affect any part of the gastrointestinal tract, whereas UC involves only rectum and colon.

UC is a chronic idiopathic inflammatory disease characterized by relapsing and remitting mucosal inflammation involving the colon and the rectum. The peak age of disease onset is between ages 30 years and 40 years. Although the exact etiology of UC remains uncertain, a combination of patient's immune response, genetics, microbiome, and environment plays an important role in the development of the inflammation. The incidence of UC is similarly in men and women, but varies with ethnicity. UC has the highest incidence in the USA, UK and Sweden. In Egypt, the prevalence is low, but newly diagnosed cases are increasing rapidly.

The most common signs and symptoms of UC include bloody stool, diarrhea, vomiting, fatigue, abdominal pain, fever, weight loss with enhanced risk of colorectal cancer and several extra intestinal manifestations (e.g., arthritis, uveitis, and skin disease). Symptoms are often non-specific, and patients frequently suffer from long-lasting subclinical disease activity that is difficult to monitor and treat.

A chronic uncontrolled immune response is the net result of excessive immune activity of effector lymphocytes with increased production of pro-inflammatory cytokines, while regulatory immune cells and mediators fail to maintain tissue homeostasis. Chronically active inflammation is directly coupled to the generation and release by immune cells of reactive oxygen species (ROS), serving as important signaling molecules that contribute to their immunological functions. The continuous release of ROS in the local microenvironment of actively inflamed mucosal lesions causes extensive cellular and molecular damage, leading to intestinal inflammation and increased tissue destruction.

Oxidative stress which is an imbalance between ROS and antioxidant activity as the result of either ROS overproduction or a decreased antioxidant activity, has been proposed as one of the major mechanism involved in the pathophysiology of UC. Once the free radicals are formed, this reactive species begins to interact with the molecular complexes causing cellular oxidative damage. Under physiological conditions, their generation is controlled by the antioxidant system, which consists of enzymes such as superoxide dismutase (SOD), catalase, and glutathione peroxidase (GPX).

Increased ROS have destructive effects which can affect lipids, proteins, and nucleic acids that causes lipid peroxidation, enzymatic dysfunction, and DNA strand break products. These destructive effects can be removed by antioxidant balance, which acts like free radical scavengers or cellular oxidation inhibitors. The main cellular antioxidant enzymes involved in the inhibition are catalase, SOD, and GPX. Activated neutrophils and macrophages are responsible for ROS generation, and their levels can be correlated with the severity of inflammation. It has been shown that IL 1 and TNFα cytokines can be inhibited by antioxidants administered to patients with UlcerativeColitis.

The American College of Gastroenterology (ACG) recommends performing a complete blood count (CBC), and measuring inflammatory markers such as c-reactive protein (CRP), erythrocyte sedimentation rate (ESR). It also recommends measuring Liver transaminases (aspartate and alanine aminotransferase). Measurement of fecal calprotectin is useful for screening intestinal inflammation associated with disease activity.

Silymarin (milk thistle), an extract obtained from Silybum marianum seeds, is one of these natural sources containing a complex of flavonolignans with a potent intracellular antioxidant property. The first usage of Milk thistle was for its hepatoprotective and antioxidant activities, but in the recent years its benefit has been reported in control of immune based murine colitis by healing of bowel histology and reduction of bowel inflammatory cytokines especially TNF-α, interleukin-1β (IL-1β), and nuclear factor κB (NF-κB). Silymarin has numerous health benefits and exerts its effects via various molecular mechanisms. Silymarin has anti-viral, immunomodulation, anti-inflammatory effects as well as antioxidant properties by scavenging free radicals and increasing the glutathione concentrations, anti-arthritis, antidiabetic, protective and wound healing effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of both sexes aged from 18 years to 65 years.
2. Adults with normal kidney and liver functions.
3. Patients who sign the consent and willing to participate in the study.
4. Patients with UC according to American College of Gastroenterology Clinical Guidelines for diagnosis Ulcerative Colitis having clinical signs and symptoms with a completed medical workup, colonoscopy, pathological and laboratory data confirming UC

Exclusion Criteria:

1. Previous hypersensitivity or anaphylactic reaction to silymarin.
2. Significant renal and hepatic impairment.
3. Patients who refuse to participate.
4. Pregnant women, breastfeeding women and smokers.
5. Patients taking corticosteroids or biological therapy.
6. Patients taking any other antioxidants.
7. Patients having other concomitant diseases where oxidative stress is involved in the etiology such as chronic liver disease, pulmonary infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
2 points or more decrease in the Mayo score from baseline | baseline, 3 months
  The Mayo score is one of the most commonly used disease activity indices in controlled trials in UC. In its complete form, it is composed of four parts: rectal bleeding, stool frequency, physician assessment, and endoscopy appearance. Each part is rated from 0 to 3, giving a total score of 0 to 12. A score of 3 to 5 points indicates mildly active disease, a score of 6 to 10 points indicates moderately active disease, and a score of 11 to 12 points indicates severely active disease.

SECONDARY OUTCOMES:
The change in the level of fecal calprotectin | baseline, 3 months
  Significant decrease in the marker level
The change in the level of superoxide dismutase | baseline, 3 months
  Significant decrease in the marker level
The change in the level of TNF-α. | baseline, 3 months
  Significant decrease in the marker level

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M Ghobashy ElHaggar, Professor, Study Director — Tanta University; Hussein A ElAmin Hammam, Professor, Study Director — Assiut University; Dalia R Mohammed ElAfify, Asst.Prof, Study Chair — Tanta University
Locations (2):
- Egypt (2):
  - Mabarra Hospital, Asyut
  - Rajhy Hospital, Asyut

REFERENCES:
- See also: A comparative study of curcumin-loaded lipid-based nanocarriers in the treatment of inflammatory bowel disease — https://doi.org/10.1016/j.colsurfb.2016.03.038
- See also: Inflammatory bowel disease: cause and immunobiology — https://doi.org/10.1016/S0140-6736(07)60750-8
- See also: Clinical epidemiology of inflammatory bowel disease: incidence, prevalence, and environmental influences — https://doi.org/10.1053/j.gastro.2004.01.063
- See also: A decade of inflammatory bowel disease: a single center experience in Egypt — https://doi.org/10.1186/s43162-022-00115-x
- See also: ACG Clinical Guideline: Ulcerative Colitis in Adults — http://doi.org/10.14309/ajg.0000000000000152
- See also: British Society of Gastroenterology consensus guidelines on the management of inflammatory bowel disease in adults — https://doi.org/10.1136/gutjnl-2019-318484
- See also: Effect of silymarin on kidneys of rats suffering from alloxan-induced diabetes mellitus — https://doi.org/10.1016/j.phymed.2010.04.011
- See also: A Meta-Analysis of the Placebo Rates of Remission and Response in Clinical Trials of Active Ulcerative Colitis — https://doi.org/10.1053/j.gastro.2006.12.037
- See also: A randomized, double blinded, placebo-controlled clinical trial of silymarin in ulcerative colitis — https://doi.org/10.1007/s11655-012-1026-x